CLINICAL TRIAL: NCT01503216
Title: Safety and Bioefficacy of Vitamin D2 and Vitamin D3: Randomized Trial With Human Volunteers
Brief Title: Safety and Bioefficacy of Vitamin D2 and Vitamin D3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulrike Lehmann (Other)
Responsible Party: Sponsor-Investigator, Ulrike Lehmann, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMBF 0315668A
Record Dates: First submitted 2011-10-24; First posted 2012-01-02 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Vitamin D Deficiency
Keywords: randomized controlled trial; vitamin D; bioavailability
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cholecalciferol (Experimental): Human volunteers receiving cholecalciferol (vitamin D3) for 8 weeks
  Interventions: Dietary Supplement: cholecalciferol
- Ergocalciferol (Experimental): Ergocalciferol 2000 IU per day for 8 weeks
  Interventions: Dietary Supplement: ergocalciferol
- Placebo (Placebo Comparator): Placebo for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — cholecalciferol, 2000 IU per day, 8 weeks
  Other Names: Cholecalciferol, vitamin D3
  Arms: cholecalciferol
Dietary Supplement: ergocalciferol — vitamin d2, 2000 IU per day for 8 weeks
  Arms: Ergocalciferol
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the bioavailability of vitamin D2 and D3 as measured by the increase of the specific hydroxy forms in serum (25(OH)D2 and 25(OH)D3, respectively, and by total 25(OH)D.

DETAILED DESCRIPTION:
Study design: Human volunteers will receive supplements containing either vitamin D2 or D3 for a period of 8 weeks. At baseline, after 4 weeks and after 8 weeks, 25(OH)D2, 25(OH)D3 and total 25(OH)D will be measured in serum as the main outcome variables. Additional outcome variables are the Ca concentration in serum, PTH concentration in serum, ambulatory blood pressure and heart rate, and renin expression in peripheral mononuclear cells.

Groups/Cohorts Assigned Interventions

1. Placebo group
2. Vitamin D2-group Daily treatment with vitamin d2-supplements (containing 2000 IU per capsule)
3. Vitamin D3-group Daily treatment with vitamin d3-supplements (containing 2000 IU per capsule)

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* healthy

Exclusion Criteria:

* supplementation of vitamin d and calcium
* hypercalcemia
* hypercalciuria
* chronical illness (diabetes, kidney diseases, cardiovascular diseases)
* serum-creatinine above 115 mmol/l
* pregnancy or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
change of 25-hydroxvitamin D | after 4 and 8 weeks of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Jutta Dierkes, Prof. Dr., Study Director — Institut für Agrar- und Ernährungswissenschaften

REFERENCES:
- [Derived] Lehmann U, Hirche F, Stangl GI, Hinz K, Westphal S, Dierkes J. Bioavailability of vitamin D(2) and D(3) in healthy volunteers, a randomized placebo-controlled trial. J Clin Endocrinol Metab. 2013 Nov;98(11):4339-45. doi: 10.1210/jc.2012-4287. Epub 2013 Sep 3. PMID 24001747